CLINICAL TRIAL: NCT00053534
Title: Heart Failure in the Community
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1207; R01HL072435 (NIH)
Record Dates: First submitted 2003-01-30; First posted 2003-01-31 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-02

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Heart Failure; Coronary Disease; Diabetes Mellitus; Hypertension; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Heart Failure; Coronary Disease; Diabetes Mellitus; Hypertension; Obesity

SUMMARY:
To monitor trends in congestive heart failure in Olmsted County, Minnesota.

DETAILED DESCRIPTION:
BACKGROUND:

Heart failure (HF) is designated as an emerging epidemic. Yet, it is not fully characterized. Most data, derived from hospital discharges, cannot measure incidence, have uncertain validity and cannot capture the full burden of heart failure because of the shift towards outpatient care. Regarding its etiology, the respective role of hypertension and coronary heart disease (CHD) is controversial. Moreover, the prevalence of obesity and diabetes mellitus is increasing, both conditions linked to heart failure via several mechanisms such that their contribution to heart failure could conceivably be increasing but remains to be examined. Finally, while the existence of diastolic heart failure is recognized, its diagnosis is exclusionary based on symptoms of heart failure in the absence of left ventricular systolic dysfunction. This approach is unsatisfactory, thus the contribution of diastolic heart failure to heart failure remains contentious. These striking gaps in knowledge underscore the necessity of a rigorous investigation of the heart failure epidemic. Through surveillance of the Olmsted County community, previous studies have demonstrated the postponement of coronary heart disease towards older ages and the decline over time in the severity of hospitalized myocardial infarction and the incidence of heart failure after myocardial infarction. This implies that, if coronary heart disease is the main cause of heart failure, heart failure should be postponed towards older ages and its incidence rate relatively stable. During the same period, preliminary findings on heart failure surveillance suggest that the incidence of first clinical diagnosis of heart failure may not be increasing as much as implied by hospital discharges and that adverse trends may be occurring preferentially among younger ages. These data from the same community are challenging to reconcile with the concept of an ongoing major contribution of coronary heart disease to an epidemic of heart failure, thereby underscoring the need to rigorously study the epidemiology of heart failure.

DESIGN NARRATIVE:

The study has three specific aims and uses a community surveillance approach which is integrated with ongoing work on coronary heart disease surveillance to investigate the heart failure epidemic in Olmsted County by characterizing its magnitude and determinants and studying prospectively the contribution of diastolic heart failure. Aim 1 will estimate the secular trends in the incidence and in the outcome of validated heart failure to test the hypotheses that there has been an increase in the incidence of heart failure, which differs by age and sex and that the survival of heart failure improved while hospitalization for heart failure has increased. Aim 2 will use a case-control approach to characterize the etiology of heart failure and its changes over time and to test the hypotheses that coronary heart disease and hypertension confer an excess risk of heart failure, the magnitude of which is declining over time, that obesity and diabetes mellitus confer an excess risk of heart failure the magnitude of which is increasing and that the population attributable risk of coronary heart disease and hypertension for heart failure is declining, while that of obesity and diabetes mellitus is increasing over time. Aim 3 will prospectively characterize the contribution of diastolic heart failure to heart failure using brain natriuretic peptide (BNP) among persons with heart failure and define the prognostic value of BNP in all cases of heart failure.

ELIGIBILITY:
No eligibility criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-01; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Veronique Roger — Mayo Clinic

REFERENCES:
- [Background] Bursi F, Enriquez-Sarano M, Nkomo VT, Jacobsen SJ, Weston SA, Meverden RA, Roger VL. Heart failure and death after myocardial infarction in the community: the emerging role of mitral regurgitation. Circulation. 2005 Jan 25;111(3):295-301. doi: 10.1161/01.CIR.0000151097.30779.04. Epub 2005 Jan 17. PMID 15655133
- [Background] Roger VL, Weston SA, Redfield MM, Hellermann-Homan JP, Killian J, Yawn BP, Jacobsen SJ. Trends in heart failure incidence and survival in a community-based population. JAMA. 2004 Jul 21;292(3):344-50. doi: 10.1001/jama.292.3.344. PMID 15265849
- [Background] Pakhomov SV, Buntrock J, Chute CG. Prospective recruitment of patients with congestive heart failure using an ad-hoc binary classifier. J Biomed Inform. 2005 Apr;38(2):145-53. doi: 10.1016/j.jbi.2004.11.016. PMID 15797003